CLINICAL TRIAL: NCT02069548
Title: Analysis of 3-D Movements of the Head in Cervical Dystonia: Comparative Assessment of the Cervical Mobility With the Mean of 3D Sensors Motion Capture Between Patients With Cervical Dystonia and Control Subjects
Brief Title: Analysis of Three-dimensional Movements of the Head in Cervical Dystonia
Acronym: STAC1
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-A01400-45
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical dystonia
- matched controlled subjects: matched in age (+/- 5 years) and gender

SUMMARY:
This study addresses postures and range of motion in cervical dystonia (Spasmodic Torticollis). It uses 3D miniature and wireless motion captures sensors, and aims to increase the understanding of the biomechanics of the movement disorders of the cervical column in this pathology. In addition, the clinical state of cervical dystonia of the patients will be assessed, using the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS). The investigators will compare the results between control and study groups.

ELIGIBILITY:
Inclusion Criteria:

* Segmental cervical dystonia diagnosed by a neurological specialist in movement disorders

Exclusion Criteria:

* Neurological pathology other than cervical dystonia such as Parkinson's disease, head tremor, severe pain or cervical ailment, which would have required a treatment within the last six months
* Neuroleptic treatment in course
* Pregnancy
* breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study-group: 30 patients meeting the criteria for cervical dystonia (Spasmodic Torticollis) and without botulinum toxin injections during the last 6 previous months before baseline. Patients will be selected consecutively among the outpatients with movement disorder of 3 study sites: Fondation OPH Rothschild, Salpetriere Hospital and Sainte-Anne Hospital (Paris)
  Control-group: 30 healthy volunteers matched in age (+/- 5 years) and gender with the 30 CD subjects. They will be selected in Sainte-Anne Hospital (Paris)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Range of motion of the voluntary mobility of the cervical spine in the three spatial planes | baseline
  Range of motion of the voluntary mobility of the cervical spine in the three spatial planes, measured in patients and matched control subjects

SECONDARY OUTCOMES:
movements disorders in cervical dystonia | baseline
  correlations between the movements disorders (range of motion, angular velocity, direction deviation) and the clinical characteristics of cervical dystonia, among patients with cervical dystonia
head posture | baseline
  influence of vision on the head posture
range of motion | baseline
  influence of vision on the range of motion

OTHER OUTCOMES:
score on the Toronto Western Spasmodic torticolis rating scale | baseline
  clinical characteristics of cervical dystonia

CONTACTS AND LOCATIONS:
Overall Officials: Sangla Sophie, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France